CLINICAL TRIAL: NCT04332822
Title: R-MINI-CHOP Versus R-MINI-CHP in Combination With Polatuzumab-vedotin, as Primary Treatment for Patients With Diffuse Large B-cell Lymphoma, ≥80 Years, or Frail ≥75 Years - an Open Label Randomized Nordic Lymphoma Group Phase III Trial
Brief Title: A Randomized, Multicenter, Phase III Trial Comparing Treatment With R-mini-CHOP With R-mini-CHP + Polatuzumab Vedotin in Patients With Diffuse Large Cell B Cell Lymphoma
Acronym: POLAR BEAR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nordic Lymphoma Group (Network)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NLG-LBC7 POLAR BEAR
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-02

CONDITIONS: DLBCL; Diffuse Large B Cell Lymphoma
Keywords: DLBCL; Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - R-mini-CHOP (Active Comparator): Cycles 1-6, duration 21 days
  * Rituximab 375 mg/m2 i.v., day 1, cycle 1. 1400 mg s c OR 375 mg/m2 i. v. cycles 2-6
  * Cyclophosphamide 400 mg/m2 i.v., day 1, cycles 1-6
  * Doxorubicin 25 mg/m2 i.v., day 1, cycles 1-6
  * Vincristine 1 mg i.v. (total dose), day 1, cycles 1-6
  * Prednisone, 40 mg/m2 p.o, days 1-5, , cycles 1-6
  Interventions: Drug: R-mini-CHOP
- Arm B - R-pola-mini-CHP (Experimental): Cycles 1-6, duration 21 days
  * Rituximab 375 mg/m2 i.v., day 1, cycle 1. 1400 mg s c OR 375 mg/m2 i. v. cycles 2-6
  * Cyclophosphamide 400 mg/m2 i.v., day 1, cycles 1-6
  * Doxorubicin 25 mg/m2 i.v., day 1, cycles 1-6
  * Prednisone, 40 mg/m2 p.o, days 1-5, , cycles 1-6
  * Polatuzumab vedotin 1.8 mg/kg i.v day 1 cycles 1-6
  Interventions: Drug: R-pola-mini-CHP

INTERVENTIONS:
Drug: R-pola-mini-CHP — * Rituximab 375 mg/m2 iv, day 1, cycle 1. 1400 mg s c OR 375 mg/m2 iv cycles 2-6
  * Cyclophosphamide 400 mg/m2 iv, day 1, cycles 1-6
  * Doxorubicin 25 mg/m2 iv , day 1, cycles 1-6
  * Prednisone, 40 mg/m2 po, days 1-5, cycles 1-6 - round up to nearest 25 mg
  * Polatuzumab vedotin 1.8 mg/kg iv day 1 cycles 1-6
  Arms: Arm B - R-pola-mini-CHP
Drug: R-mini-CHOP — * Rituximab 375 mg/m2 i.v., day 1, cycle 1. 1400 mg s c OR 375 mg/m2 i. v. cycles 2-6
  * Cyclophosphamide 400 mg/m2 i.v., day 1, cycles 1-6
  * Doxorubicin 25 mg/m2 i.v., day 1, cycles 1-6
  * Vincristine 1 mg i.v. (total dose), day 1, cycles 1-6
  * Prednisone, 40 mg/m2 p.o, days 1-5, , cycles 1-6
  Arms: Arm A - R-mini-CHOP

SUMMARY:
This is a phase III, randomized, open-label, multicenter trial, conducted in Sweden, Norway, Finland, Denmark, Italy, Australia and New Zealand, in elderly patients with untreated diffuse large B-cell lymphoma. Elderly is defined as either ≥80 years of age, or ≥75 years and frail, according to a simplified Comprehensive Geriatric Assessment. Patients will be randomized 1:1 to either the standard treatment for this population, R-miniCHOP, or an experimental regimen, R-pola-miniCHP, where vincristine is substituted by an immunoconjugate, polatuzumab vedotin. The duration of the screening period is up to 4 weeks. The duration of active treatment is 18 weeks in both arms, and patients will be followed up to 36 months after end of treatment. Start of enrollment is planned in Q1 2020, and the last visit of the last patient included (end of trial) is estimated in Q1 2027.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥80 years or frail ≥75 years, according to simplified comprehensive geriatric assessment
* Histologically confirmed lymphoma belonging to one of the following subtypes:

  1. diffuse large B-cell lymphoma, including transformation from an indolent lymphoma
  2. follicular lymphoma grade 3B
  3. T-cell/histiocyte-rich LBCL
  4. primary cutaneous DLBCL, leg type
  5. EBV-positive DLBCL, NOS
  6. primary mediastinal LBCL
  7. high grade B-cell lymphoma with MYC/BCL2 rearrangement
* Stage II-IV disease
* At least 1 measurable site of disease (>1.5 cm long axis)
* No previous treatment for lymphoma
* WHO performance status 0 - 3 (Grade 3 if related to DLBCL)
* Written informed consent

Exclusion Criteria:

* Severe cardiac disease: NYHA grade 3-4
* CNS involvement at diagnosis
* Uncontrolled serious infection
* Impaired liver (transaminases > 3x normal upper limit or bilirubin > 1.5 x normal upper limit, unless due to Gilbert´s syndrome) , renal (GFR<30ml/min) or other organ function not caused by lymphoma, which will interfere with the treatment.
* Absolute neutrophil count (ANC) <1000 cells/µL or platelets <100,000 cells/µL, unless due to lymphoma
* Any other prior malignancy than non-melanoma skin cancer or stage 0 (in situ) cervical carcinoma, unless treated with curative intent, and without relapse since 2 years, or low grade prostate cancer, not in need of treatment
* Psychiatric illness or condition which could interfere with their ability to understand the requirements of the study
* Known hypersensitivity to rituximab, polatuzumab vedotin, cyclophosphamide, vincristine or doxorubicin, or HACA against rituximab
* Peripheral neuropathy grade ≥ 2

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-08-19 (Actual); Primary Completion 2025-12-28 (Estimated); Study Completion 2028-12-28 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS). | 2 years.
  Interval between randomization date and date of documented progression, first relapse, or death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Mats Jerkeman, Principal Investigator — Department of Oncology, Skåne University Hospital
Locations (69):
- Australia (21):
  - Border Medical Oncology Research Unit, Albury
  - Royal Prince Alfred Hospital, Camperdown
  - Coffs Harbour, Coffs Harbour
  - Concord Repatriation General Hospital, Concord
  - Tweed Valley Hospital, Cudgen
  - The Canberra Hospital, Garran
  - Royal Hobart Hospital, Hobart
  - Liverpool, Liverpool
  - Bendigo, Melbourne
  - Northern Health, Melbourne
  - St Vincent's Hospital Melbourne, Melbourne
  - Western Health, Melbourne
  - Fiona Stanley Hospital, Murdoch
  - Orange Health, Orange
  - Royal Perth Hospital, Perth
  - Port Macquarie, Port Macquarie
  - Prince of Wales Hospital, Randwick
  - Royal North Shore Hospital, St Leonards
  - Sunshine Coast University Hospital, Sunshine Coast
  - Calvary Mater Newcastle, Waratah
  - Westmead, Westmead
- Denmark (8):
  - Department og Hematology, Aalborg University Hospital, Aalborg
  - Department of Hematology, Aarhus University Hospital, Aarhus
  - Clinic of Hematology L-4241, Rigshospitalet, Copenhagen
  - Sydvestjysk Sygehus, Esbjerg
  - Regionshospitalet Holstebro, Holstebro
  - Department of Hematology X, Odense University Hospital, Odense
  - Department of Hematology, Zeeland University Hospital Roskilde, Roskilde
  - Vejle Sygehus, Vejle
- Finland (5):
  - Department of Hematology, Helsinki University Hospital Comprehensive Cancer Center, Helsinki
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- Italy (12):
  - Centro di riferimento oncologico di Aviano, Aviano
  - Istituto Tumori "Giovanni Paolo II" I.R.C.C.S Bari, Bari
  - The G.O.M. Bianchi-Melacrino-Morelli in Reggio Calabria, Calabria
  - Ospedale San Gerardo di Monza, Monza
  - Azienda Ospedaliera Univeristaria Federico II di Napoli, Napoli
  - Istituto Nazionale Tumori "Fondazione Pascale" Napoli, Napoli
  - Azienda Ospedaliera San Camillo Forlanini di Roma, Roma
  - IRCCS San Raffaele Scientific Institute, Segrate
  - Azienda Sanitaria Universitaria Integrata di Trieste, Trieste
  - AOU San Luigi Gonzaga - Orbassano University of Turin, Turin
  - Azienda Sanitaria Universitaria Integrata di Udine, Udine
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- New Zealand (2):
  - Auckland City Hospital, Grafton
  - Wellington Blood and Cancer Centre, Wellington
- Norway (8):
  - Haukeland Universitetshospital, Bergen
  - Kalnes Hospital (Østfold), Grålum
  - Sykehuset Innlandet, Innlandet
  - Akershus University Hospital, Oslo
  - Avd. for Kreftbehandling, Oslo universitetssykehus, Oslo
  - Avdeling for Blod- og Kreftsykdommer, Stavanger Universitetssykehus, Stavanger
  - Kreftklinikken, St Olavs Hospital, Trondheim
  - Sykehuset i Vestfold, Tønsberg
- Sweden (13):
  - Medicinkliniken, Södra Älvsborg Sjukhus, Borås
  - Department of Hematology and Coagulation, Sahlgrenska University Hospital, Gothenburg
  - Department of Medicine, Halmstad Country Hospital, Halmstad
  - Department of Internal Medicine, Kalmar County Hospital, Kalmar
  - Hematologiska Kliniken, Universitetssjukhuset, Linköping
  - Department of Oncology, Skåne University Hospital, Lund
  - Department of Oncology, Örebro University Hospital, Örebro
  - Department of Medicine, Sunderbyn Hospital, Södra Sunderbyn
  - Center of Hematology, Karolinska University Hospital, Stockholm
  - Uddevalla Sjukhus, Uddevalla
  - Cancercentrum, Norrlands universitetsjukhus, Umeå
  - Department of Oncology, Uppsala Academic Hospital, Uppsala
  - Varberg Hospital, Varberg